CLINICAL TRIAL: NCT01780571
Title: Continuous Positive Airway Pressure/Pressure Support Preoxygenation of Morbidly Obese Patients
Brief Title: CPAP/PSV Preoxygenation in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Näslund, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KIDS CPAP
Record Dates: First submitted 2012-12-09; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Anaesthesia
Keywords: Obesity; general anaesthesia; preoxygenation; atelectasis
MeSH Terms: conditions — Obesity; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Neutral pressure breathing after 2 min preoxygenation
- Active group (Active Comparator): CPAP 5cm H2O + PSV 5cm H2O breathing after 2 min preoxygenation
  Interventions: Procedure: CPAP 5 cm H2O + PSV 5 cm H2O

INTERVENTIONS:
Procedure: CPAP 5 cm H2O + PSV 5 cm H2O — Patients in the intervention group received Continuous Positive Airway Pressure (5 cm H2O) and Pressure Supported Ventilation (5 cm H2O)
  Arms: Active group

SUMMARY:
The purpose of this study is to determine whether continuouse positive airway pressure (CPAP), during induction of anaesthesia in morbidly obese patients, result in higher levels of oxygen in the blood.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) > 35 kg/m2
* scheduled to undergo elective gastric bypass surgery
* age ≥ 18 years
* ASA Physical Status Classification II-III

Exclusion Criteria:

* significant cardiopulmonary disease
* previous abdominal or thoracic surgery
* inability to comprehend the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Post intubation PaO2levels | 5 minutes after intubation
  PaO2 levels is measured within 5 minutes after the completion of intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Danderyd Hospital, Stockholm, Sweden